CLINICAL TRIAL: NCT02284880
Title: Comparative Bioavailability Study of Two Different Sources of Eslicarbazepine Acetate in Healthy Subjects
Brief Title: Comparative Bioavailability Study of Two Different Sources of Eslicarbazepine Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIA-2093-130
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 BIA 2-093 (Experimental): Subjects randomly received on period 1 and 2, either a single 400 mg tablet of ESL (MF - marketed formulation), or a single 400 mg tablet of ESL (TBM - o-be-marketed);
  Interventions: Drug: BIA 2-093
- Group 2 BIA 2-093 (Experimental): Subjects randomly received on period 1 and 2, either a single 800 mg tablet of ESL (MF - marketed formulation), or a single 800 mg dose of ESL (TBM - o-be-marketed).
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093 — MF - Marketed formulation
  Other Names: ESL, Eslicarbazepine acetate
Drug: BIA 2-093 — TBM - to-be-marketed
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
Phase I, two-centre, open-label, randomized, gender-balanced, single-dose, laboratory blinded, two-period, two-sequence, crossover study in 2 groups of 20 healthy male and female subjects, to demonstrate the bioequivalence (BE) between two active product ingredient (API) sources of eslicarbazepine acetate (ESL)

DETAILED DESCRIPTION:
Phase I, two-centre, open-label, randomized, gender-balanced, single-dose, laboratory blinded, two-period, two-sequence, crossover study in 2 groups of 20 healthy male and female subjects. The study consisted in 2 periods separated by a wash-out of at least 7 days between doses. To demonstrate the bioequivalence (BE) between two active product ingredient (API) sources [current API source - marketed formulation (MF) versus new API source - to-be-marketed (TBM)] of eslicarbazepine acetate (ESL)

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form before any study-specific screening procedure was performed,
* Healthy male or female 18 to 55 of age, inclusive,
* Had a BMI within the range of 18 to 25 kg/m2 inclusive at screening,
* Had a physical examination, vital signs, electrocardiogram (ECG) and routine laboratory tests within normal ranges or considered as non clinically significant (NCS) by the Investigator,
* Non-smokers or smokers of less than 10 cigarettes per day,
* If female, she was not of childbearing potential by reason of surgery (hysterectomy, bilateral oophorectomy or tubal ligation) or, if of childbearing potential, she had to be using one of the following effective method of contraception (intrauterine device (IUD) or abstention or condom) for the duration of the trial and had to have a negative urine pregnancy test at screening visit and upon each admission period.

Exclusion Criteria:

* Had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue disease or disorders, or have a clinically relevant surgical history,
* Presented any disease or condition (medical or surgical) which, in the opinion of the Investigator, that may have interfered with the absorption, distribution, metabolism or excretion of study drug,
* Had a history of relevant atopy or any drug hypersensitivity (including known hypersensitivity to eslicarbazepine acetate or any of its excipients),
* Had a history of alcoholism or drug abuse within 1 year before D 1,
* Consumption of more than 50 g of ethanol per day (12.5 Centiliters [cL] glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g),
* Use of medicines within 2 weeks of admission to first treatment period that could affect, in the Investigator's opinion, the safety of the subject,
* Had used any investigational drug or participated in any clinical trial within 2 months of admission to first treatment period,
* Had donated or received any blood or blood products within 2 months prior to screening,
* Could not communicate reliably with the investigator, was unlikely to co-operate with the requirements of the study,
* Was unwilling or unable to give written informed consent,
* If female, was pregnant or breast-feeding,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- 400 mg BIA 2-093 Group 1; 800 mg BIA 2-093 Group 1: In Group 1, subjects received on period 1 and 2: 400 mg BIA 2-093 ESL: MF first, then TBM
- 400 mg BIA 2-093 Group 2; 800 mg BIA 2-093 Group 2: In Group 2, subjects received on period 1 and 2: 400 mg BIA 2-093 ESL: TBM first, then MF
Period: Overall Study
Arm/Group | 400 mg BIA 2-093 Group 1 | 400 mg BIA 2-093 Group 2 | 800 mg BIA 2-093 Group 1 | 800 mg BIA 2-093 Group 2
Started | 11 | 9 | 10 | 10
First Period (4 Days) | 11 | 9 | 10 | 10
Wash-out Period (7 Days) | 11 | 9 | 10 | 10
Second Period (4 Days) | 11 | 9 | 8 | 10
Completed | 11 | 9 | 8 | 10
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- 400 mg BIA 2-093: In Group 1, subjects received randomly on period 1 and 2, either a single 400 mg tablet of ESL (MF), or a single 400 mg tablet of ESL (TBM).
- 800 mg BIA 2-093: In Group 2, subjects received randomly on period 1 and period 2, either a single 800 mg tablet of ESL (MF), or a single 800 mg dose of ESL (TBM).
- Total: Total of all reporting groups
Arm/Group | 400 mg BIA 2-093 | 800 mg BIA 2-093 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration
Description: Reference - MF - marketed formulation Test - TBM - to-be-marketed BIA 2-005 - BIA 2-093 metabolite
Time Frame: pre-dose then 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose on each dosing period
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 400 mg BIA 2-093 | 800 mg BIA 2-093
Number analyzed (Participants) | 20 | 18
ng/ml
  Cmax (BIA 2-005 Reference) | 6461 (1346) | 13183 (2564)
  Cmax (BIA 2-005 Test) | 6547 (1524) | 12988 (2215)

2. Primary Outcome: Tmax - Time of Occurrence of Cmax
Description: Reference - MF - marketed formulation Test - TBM - to-be-marketed
  BIA 2-005 - BIA 2-093 metabolite
Time Frame: pre-dose then 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose on each dosing period
Measure: Median (Full Range); unit: hours
Arm/Group | 400 mg BIA 2-093 | 800 mg BIA 2-093
Number analyzed (Participants) | 20 | 18
hours
  Tmax (BIA 2-005 Reference) | 2.00 [0.50 to 6.00] | 2.00 [1.00 to 4.02]
  Tmax (BIA 2-005 Test) | 2.00 [0.50 to 6.00] | 1.75 [1.00 to 6.00]

3. Primary Outcome: AUC0-t - Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to the Last Sampling Time at Which Concentrations Were at or Above the Limit of Quantification
Description: Reference - MF - marketed formulation Test - TBM - to-be-marketed
  BIA 2-005 - BIA 2-093 metabolite
Time Frame: pre-dose then 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose on each dosing period
Measure: Mean (Standard Deviation); unit: ng.hr/ml
Arm/Group | 400 mg BIA 2-093 | 800 mg BIA 2-093
Number analyzed (Participants) | 20 | 18
ng.hr/ml
  AUC0-t (BIA 2-005 Reference) | 112568 (23011) | 279035 (60183)
  AUC0-t (BIA 2-005 Test) | 108224 (23971) | 278734 (61738)

ADVERSE EVENTS:
Groups:
- Before Treatment: Before treatment with ESL ESL - Eslicarbazepine acetate, BIA 2-093
- 400 mg Tablet of ESL (MF): 400 mg tablet of ESL (MF) ESL - Eslicarbazepine acetate, BIA 2-093 MF - Marketed formulation
- 400 mg Tablet of ESL (TBM): 400 mg tablet of ESL (TBM) ESL - Eslicarbazepine acetate, BIA 2-093 TBM - To be marketed
- 800 mg Tablet of ESL (MF): 800 mg tablet of ESL (MF) ESL - Eslicarbazepine acetate, BIA 2-093 MF - Marketed formulation
- 800 mg Tablet of ESL (TBM): 800 mg tablet of ESL (TBM) ESL - Eslicarbazepine acetate, BIA 2-093 TBM - To be marketed
- After Follow-up Visit: After Follow-up visit ESL - Eslicarbazepine acetate, BIA 2-093 MF - Marketed formulation TBM - To be marketed
Arm/Group | Before Treatment | 400 mg Tablet of ESL (MF) | 400 mg Tablet of ESL (TBM) | 800 mg Tablet of ESL (MF) | 800 mg Tablet of ESL (TBM) | After Follow-up Visit
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20 | 0/20 | 0/20 | 0/18 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 0/20 | 1/20 | 4/20 | 4/18 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Before Treatment (N=40) | 400 mg Tablet of ESL (MF) (N=20) | 400 mg Tablet of ESL (TBM) (N=20) | 800 mg Tablet of ESL (MF) (N=20) | 800 mg Tablet of ESL (TBM) (N=18) | After Follow-up Visit (N=40)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other